CLINICAL TRIAL: NCT05698524
Title: A Phase I Study of Metronomic Temozolomide With Abexinostat (PCI-24781) for Patients With Recurrent High Grade Glioma
Brief Title: A Study of Temodar With Abexinostat (PCI-24781) for Patients With Recurrent Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0809-22-FB
Record Dates: First submitted 2022-12-20; First posted 2023-01-26 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Recurrent High Grade Glioma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma | interventions — abexinostat; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Participants will receive a combination of PCI-24781/Abexinostat and temozolomide: loading dose of PCI-24781/Abexinostat prior to the start of Cycle 1, PCI-24781/Abexinostat by mouth twice a day starting 7 days prior to Cycle 1, Day 1 and ending 4 days prior to Cycle 1, Day 1.
  Participants will continue taking PCI-24781/Abexinostat on days 1 - 4, 8 - 11, and 15 - 18 of each 28 day cycle, starting with Cycle 1, Day 1. The initial dose level is 60 mg of PCI-2478/Abexinostat by mouth twice daily. The dose level may be escalated based on results of interim data analysis.
  Participants will additionally initiate metronomic temozolomide on Cycle 1, Day 1 at a dose of 50 mg/m2, taken by mouth twice daily and continue the PCI-24781/Abexinostat and metronomic temozolomide regimen until disease progression or intolerance.
  Interventions: Drug: PCI 24781; Drug: Temozolomide

INTERVENTIONS:
Drug: PCI 24781 — Participants will take PCI-24781/Abexinostat on days 1 - 4, 8 - 11, and 15 - 18 of each 28-day cycle.
  Other Names: Abexinostat
Drug: Temozolomide — Participants will receive temozolomide at a dose of 50 mg/mg2, taken by mouth once daily.
  Other Names: Temodar

SUMMARY:
Glioblastoma (GBM), WHO grade IV glioma, represents the majority of adult malignant primary brain tumors, with an incidence of 2-3 per 100,000 person-years. The survival for GBM has increased in the last decade but is still low with a median survival of 15-18 months. Recurrence after initial standard therapy, radiation therapy and chemotherapy with temozolomide, few options are available. Even with further therapy, median progression free survival at 6 months after first relapse (PFS-6) is only 15%. Similarly, anaplastic astrocytoma and anaplastic oligodendroglioma, grade III gliomas, once recurrent after radiation therapy and first-line chemotherapy, have identical therapeutic options and poor outcomes with PFS-6 of 31%. Temozolomide (TMZ) has a favorable side effect profile and is available orally, however, cytotoxicity occurs. Metronomic temozolomide at low doses on a continuous schedule, have demonstrated better survival in studies. This study will determine the recommended dose and the side effects of PCI-24781/Abexinostat with metronomic temozolomide.

DETAILED DESCRIPTION:
Glioblastoma (GBM), WHO grade IV glioma, represents the majority of adult malignant primary brain tumors, with an incidence of 2-3 per 100,000 person-years. The survival for GBM has increased in the last decade but is still low with a median survival of 15-18 months. Recurrence after initial standard therapy, radiation therapy and chemotherapy with temozolomide, few options are available. Even with further therapy, median progression free survival at 6 months after first relapse (PFS-6) is only 15%. Similarly, anaplastic astrocytoma and anaplastic oligodendroglioma, grade III gliomas, once recurrent after radiation therapy and first-line chemotherapy, have identical therapeutic options and poor outcomes with PFS-6 of 31%. Temozolomide (TMZ) has a favorable side effect profile and is available orally, however, cytotoxicity occurs. Metronomic temozolomide at low doses on a continuous schedule, have demonstrated better survival in studies.

Participants will be enrolled to one of each of four dose levels in cohorts of 3. Dose level escalation/de-escalation will follow Bayesian Optimal Interval (BOIN) design rules based on analysis of dose-limiting toxicities (DLTs) that occur within the first cycle of protocol treatment. Protocol treatment will continue until disease progression or intolerable toxicity. Dose Levels: 1 - 60 mg PCI-24781/Abexinostat two times daily (BID), 1.5 - 80 mg PCI-24781/Abexinostat BID, 2 - 100 mg PCI-24781/Abexinostat BID, and 3 - 140 mg PCI-24781/Abexinostat BID.

The primary study objective is to evaluate the toxicities and determine the recommended dose of PCI-24781/Abexinostat with metronomic temozolomide in participants with recurrent high grade glioma, [grade III or IV glioma (glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma)]. Other objects are to evaluate changes in the acetylation of peripheral blood mononuclear cell (PBMC) histones H3 and H4 during treatment, evaluate acetylation of histones H3 and H4 using peripheral blood exosomes, evaluate progression-free and overall survival of participants with recurrent high grade glioma treated with therapy with PCI-24781/Abexinostat and metronomic temozolomide, descriptively examine quality of life (QOL) using EORTC QLQ-C30 questionnaire and QLQ-BN20 questionnaire during treatment, characterize the pharmacokinetics (PK) of PCI-24781/Abexinostat, temozolomide, and the combination of the 2 drugs, measure tumor response, and correlate molecular profiles with tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of high grade (aka grade III or IV) glioma (anaplastic astrocytoma, anaplastic oligodendroglioma, glioblastoma, gliosarcoma)
* Prior radiation therapy and standard temozolomide; additional therapies for previous progressions are eligible (prior bevacizumab and Optune are allowed)
* Three or more months from the end of chemoradiotherapy or have biopsy or imaging consistent with disease progression
* 19 years of age or older (the age of consent in Nebraska)
* Fully recovered from any toxicity of prior therapy that, in the opinion of the investigator, could impact tolerance to the study drug
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate bone marrow reserve (ANC count ≥1,500/mm3, hemoglobin > 8 g/dL, platelet count ≥100,000/mm3)
* Adequate renal function (a serum creatinine that is at or below 2.0 mg/dL)
* Adequate hepatic function (serum AST and ALT less than 1.5 times the upper limits of normal, serum alkaline phosphatase less than 2.5 times the upper limits of normal)
* Able to provide written, informed consent
* Females of child-bearing potential must have a negative pregnancy test within 7 days of initiating study (non-child bearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)
* Females of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and up to 6 months following treatment

Exclusion Criteria:

* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of oral PCI-24781/Abexinostat, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmia, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Immunotherapy, chemotherapy, radiotherapy, corticosteroids (at dosages equivalent to prednisone > 20 mg/day) or experimental therapy (other than PCI-24781/Abexinostat PO) within 4 weeks before first dose of study drug
* Concurrent use of enzyme-inducing antiepileptic drugs (phenytoin, phenobarbital, carbamazepine, felbamate, topiramate and oxcarbazepine)
* Any other active malignancy other than nonmelanoma skin cancer or controlled prostate cancer
* Known history of Human Immunodeficiency Virus (HIV) or active infection with Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV) or any uncontrolled active systemic infection (no testing is required for eligibility)
* Creatinine > 1.5 x institutional upper limit of normal (ULN); total bilirubin > 1.5 x ULN (unless from Gilbert's disease), and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
* Pregnant or breast-feeding
* Baseline ECG duration of the ventricular action potential corrected for heart rate (QTc interval) prolongation based on Fridericia's formula is > 450 ms in males and > 470 ms in females
* Concomitant valproic acid use, or another histone deacetylases (HDAC) inhibitor
* Receiving treatment with following medications and unable to discontinue treatment or switch medications prior to study enrollment:

  * Amiodarone (Cordarone, Pacerone)
  * Arsenic trioxide (Trisenox)
  * Chlorpromazine (Aralen)
  * Cisapride (Propulsid)
  * Clarithromycin (Biaxin)
  * Disopyramide (Norpace)
  * Dofetilide (Tikosyn)
  * Doperidol (Inapsine)
  * Erythromycin (EryTab, Erythrocin)
  * Flecanide (Tambocor)
  * Haloperidol (Haldol)
  * Ibutilide (Corvert)
  * Methadone (Methadose, Dolophine)
  * Moxifloxacin (Avelox)
  * Pentamidine (Pentam, Nebupent)
  * Pimozide (Orap)
  * Procainamide (Procan, Pronestyl)
  * Quinidine (Cardioquin, Quinaglute)
  * Sotalol (Betapace)
  * Thioridazine (Mellaril)
  * Vandetanib (Zactima)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Toxicities Associated with PCI-24781/Abexinostat and Metronomic Temozolomide Therapy - Adverse Events and Serious Adverse Events | Up to 25 months
  The incidence of adverse events (AEs) and serious adverse events (SAEs) will be recorded for each dose level cohort. Toxicities will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicities will be graded on from 1 to 5, with higher numbers indicating a higher severity grade.
Toxicities Associated With PCI-24781/Abexinostat and Metronomic Temozolomide Therapy - Overall | Up to 25 months
  The frequency of overall toxicity occurrence will be categorized by toxicity grades using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicities will be graded ranging from 1 to 5, with higher numbers indicating a higher severity grade.
Recommended Dose Determination of PCI-24781/Abexinostat | Up to 20 months
  Participants who either complete the first cycle of treatment or experience a dose-limiting toxicity (DLT) within the first cycle of treatment will be considered evaluable. The target DLT rate for the maximum tolerated dose (MTD) is 0.25. The MTD determination will be based on isotonic regression. The MTD will be defined as the dose for which the isotonic estimate of the DLT rate is closest to the target DLT rate of 0.25. If a tie exists between potential doses the higher dose level will be selected when the isotonic estimate is lower than the target DLT rate and the lower dose level will be selected when the isotonic estimate is greater than or equal to the target DLT rate.
  If the observed DLT rate at the current dose is ≤ 0.197, escalate the dose to the next higher dose level. If the observed DLT rate at the current dose is > 0.298, de-escalate the dose to the next lower dose level. Otherwise, stay at the current dose level.

SECONDARY OUTCOMES:
Changes in Acetylation of Peripheral Blood Mononuclear Cell Histones, H3 and H4, During Treatment | Up to 20 months
  Peripheral blood samples collected at baseline and during treatment will be analyzed for changes in acetylation of peripheral blood mononuclear cell (PBMC) histones H3 and H4.
Changes in Acetylation of Histones, H3 and H4, Using Peripheral Blood Exosomes | Up to 20 months
  Peripheral blood samples collected at baseline and during treatment will be analyzed for changes in acetylation of peripheral blood mononuclear cell (PBMC) histones, H3 and H4, using peripheral blood exosomes.
Progression-free Survival | 36 months
  Progression-free survival (PFS), the time from treatment initiation to disease progression, will be estimated using the Kaplan-Meier method.
Overall Survival (OS) | 36 months
  Overall survival (OS), the time from treatment initiation to death from any cause, will be estimated using the Kaplan-Meier method.
Descriptive examination of patient quality of life during treatment (EORTC QLQ-C30) | 24 months
  Participant Quality of Life (QOL) will be measured throughout treatment using the European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-BN30) questionnaire. Question responses range from 1 (Not at All) to 4 (Quite a Bit). Higher scores indicate greater functioning. Two additional questions ask participants to rate overall health and quality of life using a scale ranging from 1 to 7, where higher numbers indicate more favorable outcomes.
Descriptive Examination of Participant Quality of Life During Treatment (EORTC QLQ-BN20) | 24 months
  Participant Quality of Life (QOL) will be measured throughout treatment using the European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-BN20) questionnaire. Question responses range from 1 (Not at All) to 4 (Quite a Bit). Higher scores indicate greater functioning.
Measurement of Tumor Response | Up to 36 months
  Magnetic resonance imaging (MRI) and clinical features will be used to classify tumor response as one of four categories that range from complete response to disease progression. The overall response will be assessed using Response Assessment in Neuro-Oncology (RANO) Criteria.
Correlation of Molecular Profiles With Tumor Response | Up to 36 months
  The correlation of tumor response and peripheral blood mononuclear cells (PBMC) and exosomes extracted from peripheral blood samples will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Shonka, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No